CLINICAL TRIAL: NCT05625048
Title: Urinary Incontinence After Radical Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regional Hospital West Jutland (Other)
Responsible Party: Principal Investigator, Sara Birch, Principal investigator, Regional Hospital West Jutland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-10-72-356-21
Record Dates: First submitted 2022-10-27; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Incontinence, Urinary; Radical Prostatectomy
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): The intervention group receives same treatment as the control groups and in addition transperinal ultrasound guided instruction in pelvic floor muscle training at 2nd and 3rd session.
  Interventions: Other: Transperinal ultrasound guided instruction in pelvic floor muscle training
- Control group 1 (No Intervention): The patients recieve standard care including three physiotherapist sessions; within one week preoperatively, one week postoperatively at catheter removal, and six weeks postoperatively
- Control group 2 (No Intervention): The patients recieve standard care including three physiotherapist sessions; within one week preoperatively, one week postoperatively at catheter removal, and six weeks postoperatively

INTERVENTIONS:
Other: Transperinal ultrasound guided instruction in pelvic floor muscle training — The physiotherapists uses transperinal ultrasound as a biofeedback or pedagogical tool to improve the muscle contractions and visualize the muscle work.
  Arms: Intervention group

SUMMARY:
The aims of this project are; 1) To examine the efficacy of ultrasound-guided pelvic floor muscle training compared to standard care on urinary incontinence in patients undergoing robot assisted radical prostatectomy and 2) To compare physical function, incontinence, and QoL in two groups of patients with low or high function of the pelvic floor muscles respectively before the surgery.

This study consists of two parts. The first part is a randomized controlled trial where 44 patients with weak pelvic floor muscle function are randomized to either treatment as usual (control group 1) or ultrasound-guided pelvic floor muscle training (Intervention group). In the second part the patients in control group 1 will be compared with 22 patients with normal/strong pelvic floor muscle function (control group 2).

Patients not able to perform the pelvic floor muscle test consisting of 8 repetitions of 4-seconds pelvic floor muscle contraction and 1 repetition of 15-seconds pelvic floor muscle contraction will be randomized to either intervention group or control group 1. Patients able to perform the pelvic floor muscle test will be included in control group 2.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 and above
* Diagnosis of prostatic adenocarcinoma and referred to robot assisted radical prostatectomy
* No comorbidity that prevents pelvic floor training or effects the function of the pelvic floor
* Adequacy in written and spoken Danish Performance status 0-1
* Able to understand the study procedures and willing to provide written informed consent

Exclusion Criteria:

* Major surgery within the last month that may affect pelvic floor function.
* Urinary incontinence prior to surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
24-hour pad weigh test | 12 month after the operation
  The patients have to weigh their pads before use and retain them in sealed plastic bags for repeated weight assessment when the 24-hour period has ended. The total increase in weight (gram) of all the pads will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Hospital Goedstrup, Herning, Denmark